CLINICAL TRIAL: NCT00798655
Title: A Phase II Trial of Postoperative Radiation, Cisplatin, and Panitumumab in Locally Advanced Head and Neck Cancer
Brief Title: Trial of Postoperative Radiation, Cisplatin, and Panitumumab in Locally Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Robert Ferris (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor-Investigator, Robert Ferris, Division Chief, Division Head and Neck Surgery, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-120
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Results first posted 2016-08-09 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Cancer of Head; Cancer of Head and Neck; Cancer of Neck; Cancer of the Head; Cancer of the Head and Neck; Cancer of the Neck; Head and Neck Cancer; Head Cancer; Head Neoplasms; Head, Neck Neoplasms; Neck Cancer; Neck Neoplasms; Neoplasms, Head; Neoplasms, Head and Neck; Neoplasms, Neck; Neoplasms, Upper Aerodigestive Tract; UADT Neoplasms; Upper Aerodigestive Tract Neoplasms
Keywords: panitumumab; cisplatin; radiation
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Panitumumab; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Panitumumab, Cisplatin plus radiation (Experimental): Standard radiation 60-66 Gy with 200 cGy daily fractions in 6-7 weeks Cisplatin* 30 mg/m2 IV, weekly during radiation (total of 6-7 doses based upon radiation therapy dose requirements) Panitumumab 2.5 mg/Kg IV, weekly during radiation (total of 6-7 doses based upon radiation therapy dose requirements)
  Interventions: Drug: Panitumumab; Drug: Cisplatin; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Panitumumab — Panitumumab, starting dose, 2.5mg/kg will be given as an intravenous infusion (IV) through a vein in your arm, once a week before radiation and chemotherapy for 6 weeks; treatment takes about an hour.
  The panitumumab dose will be calculated based on the subject's actual weekly body weight
  Other Names: ABX-EGF; Vectibix
Drug: Cisplatin — Cisplatin, 30 mg/m2 will be given as an intravenous infusion (IV) through a vein in your arm, once a week before radiation therapy and after panitumumab for 6 weeks; treatment takes about an hour
  Other Names: cisplatinum; cis-diamminedichloroplatinum(II); Platin
Radiation: Radiation Therapy — Radiation Therapy 60-66 Gy/200 cGy/daily, five days a week, Monday through Friday, except on weekends and holidays, for six weeks; treatments take about 20 minutes.
  Radiation will be administered either prior to chemo treatment or after chemo treatment as long as radiation is given on the same day.

SUMMARY:
The objectives for this study is as follows:

* Primary:

  * To evaluate the progression-free survival of locoregionally advanced (stages III/IV) SCCHN patients undergoing postoperative chemoradiotherapy with panitumumab.
* Secondary:

  * To evaluate the overall survival, event-free survival, and toxicities.
  * To correlate efficacy parameters with 1) EGFR and downstream pathway activation, 2) FcyR polymorphisms, and 3) serum cytokine profiles. More specifically, the aim is to demonstrate the usefulness of biomarkers (downstream signaling molecules, FcyR polymorphisms, or tumor and serum cytokine(s) in predicting progression-free survival in patients with SCCHN treated with the above treatment. Specific biomarkers that relate to Epidermal Growth Factor Receptor and angiogenesis, including EGFR, pEGFR, Src, pMAPK, pSTAT3, pSTAT5, pSTAT1, pAKT, p38, p21, p27, PARP, E-cadherin, p-ErbB3, Ki67, VEGF, and IL-8, using reverse phase protein microarrays (RPPA) will be tested in baseline archival paraffin-embedded tumor tissue. To collect tumor tissue from pretreatment biopsies for cytokine/chemokine and immune biomarker studies on tumor tissue. We plan to investigate the expression of pAKT, pMAPK, and other EGFR pathway-related markers as well angiogenesis biomarkers. In addition, EGFR polymorphisms will be studied in tumor tissue samples and serum. Additional studies may be performed in the future. Some of these studies may be performed by Amgen.

DETAILED DESCRIPTION:
Pathologically staged squamous cell carcinoma of the head and neck, stage III or IVa (AJCC 6th edition 2002) of the oral cavity, larynx, or hypopharynx that is status post potentially curative surgical resection without gross residual tumor, except the following: a)T3N0 laryngeal primary and b) any T1N1, if there are no high-risk pathologic features (high risk defined as positive margins, extracapsular spread, and perineural or angiolymphatic invasion). Patients should not have gross residual disease. No prior chemotherapy, biologic/targeted therapy (including any prior therapy which specifically and directly targets the EGFR pathway), or radiotherapy for head and neck cancer. A brief course, up to 2 weeks, of prior neoadjuvant single-agent biologic/targeted therapy of any type (except EGFR monoclonal antibodies) prior to surgical resection is permitted. No more than 7 weeks (minimum of 3 weeks) should have elapsed between surgery and initiation of radiation. No prior radiation or chemotherapy for head and neck cancer. ECOG performance status of 0-1. Patients must have normal organ and marrow function as defined below: absolute neutrophil count >=1,500/mL; Platelets >=100,000/mL; Hemoglobin >=10 g/dL; Total bilirubin 1.5 x normal institutional limits; Creatinine clearance > 60 ml/min. No prior invasive malignancy unless the DFS is 3 years or more. Age >= 18 years. Pregnant or breast-feeding women are excluded (see exclusion criteria). Informed consent must be obtained from all patients prior to beginning therapy. Patients should have the ability to understand and the willingness to sign a written informed consent document. Patients who have tumor tissue available from previous diagnostic or therapeutic procedures should submit the specimen for assessment of EGFR and related biomarkers after signing informed consent. In-Eligibility: Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements. Significant history of uncontrolled cardiac disease; i.e., uncontrolled hypertension, unstable angina, recent myocardial infarction (within prior 6 months), uncontrolled congestive heart failure, and cardiomyopathy with decreased ejection fraction. All patients will have a baseline EKG. If abnormalities consistent with active coronary artery disease are detected, the patient will be referred to a cardiologist for appropriate evaluation and management prior to treatment on study. Patients with history of hypertension must be well-controlled upon study entry (≤150/90) on a stable regimen of anti-hypertensive therapy. Patients should not have any prior history of hypertensive crisis or hypertensive encephalopathy.Patients may not be receiving any other investigational agents. No history of prior malignancy, with the exception of curatively treated squamous cell or basal carcinoma of the skin or in situ cervical cancer, or malignancy that has been treated with a curative intent with a 3-year disease-free survival. No patients with significant baseline sensory or motor neurologic deficits (> grade I neuropathy) will be treated on this study. Pregnant women are excluded from this study because chemotherapy and radiation therapy have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with chemotherapy, breastfeeding should be discontinued if the mother is treated with chemotherapy. Prior to study enrollment, women of childbearing potential (WOCBP) must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy. In addition, men enrolled on this study should understand the risks to any sexual partner of childbearing potential and should practice an effective method of birth control. All WOCBP MUST have a negative urine pregnancy test at baseline, or within 7 days prior to receiving investigational product. The minimum sensitivity of the pregnancy test must be 25 IU/L or equivalent units of HCG. If the urine pregnancy test is positive, a serum pregnancy test will then be performed to confirm the result. In the event that both the urine and serum pregnancy tests are positive, the subject must not receive investigational product and must not be enrolled in the study. In addition, all WOCBP should be instructed to contact the Investigator immediately if they suspect they might be pregnant (e.g., missed or late menstrual period) at any time during study participation. The Investigator must immediately notify Amgen in the event of a confirmed pregnancy in a patient participating in the study. Prior severe infusion reaction to a human monoclonal antibody.Prior severe infusion reaction to a human monoclonal antibody.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically staged squamous cell carcinoma of the head and neck, stage III or IVa (AJCC 6th edition 2002) of the oral cavity, larynx, or hypopharynx that is status post potentially curative surgical resection without gross residual tumor, except the following: a)T3N0 laryngeal primary and b) any T1N1, if there are no high-risk pathologic features (high risk defined as positive margins, extracapsular spread, and perineural or angiolymphatic invasion).
* Patients should not have gross residual disease.
* No prior chemotherapy, biologic/targeted therapy (including any prior therapy which specifically and directly targets the EGFR pathway), or radiotherapy for head and neck cancer. A brief course, up to 2 weeks, of prior neoadjuvant single-agent biologic/targeted therapy of any type (except EGFR monoclonal antibodies) prior to surgical resection is permitted.
* No more than 6 7 weeks (minimum of 3 weeks) should have elapsed between surgery and initiation of radiation.
* No prior radiation or chemotherapy for head and neck cancer.
* ECOG performance status of 0-1
* Patients must have normal organ and marrow function Absolute neutrophil count >/=1,500/uL Platelets >/=100,000/uL Hemoglobin >/= 10 g/dL Total bilirubin <1.5 x normal institutional limits Creatinine clearance > 60 mL/min
* No prior invasive malignancy unless the DFS is 3 years or more.
* Age > 18 years.
* Pregnant or breast-feeding women are excluded (see exclusion criteria).
* Informed consent must be obtained from all patients prior to beginning therapy. Patients should have the ability to understand and the willingness to sign a written informed consent document.
* Patients who have tumor tissue available from previous diagnostic or therapeutic procedures should submit the specimen for assessment of EGFR and related biomarkers after signing informed consent.

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements. Significant history of uncontrolled cardiac disease; i.e., uncontrolled hypertension, unstable angina, recent myocardial infarction (within prior 6 months), uncontrolled congestive heart failure, and cardiomyopathy with decreased ejection fraction. All patients will have a baseline EKG. If abnormalities consistent with active coronary artery disease are detected, the patient will be referred to a cardiologist for appropriate evaluation and management prior to treatment on study.. Patients with history of hypertension must be well-controlled upon study entry (≤150/90) on a stable regimen of anti-hypertensive therapy. Patients should not have any prior history of hypertensive crisis or hypertensive encephalopathy.
* Patients may not be receiving any other investigational agents.
* No history of prior malignancy, with the exception of curatively treated squamous cell or basal carcinoma of the skin or in situ cervical cancer, or malignancy that has been treated with a curative intent with a 3-year disease-free survival.
* No patients with significant baseline sensory or motor neurologic deficits(> grade I neuropathy) will be treated on this study.
* Pregnant women are excluded from this study because chemotherapy and radiation therapy have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with chemotherapy, breastfeeding should be discontinued if the mother is treated with chemotherapy.
* Prior to study enrollment, women of childbearing potential (WOCBP) must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy. In addition, men enrolled on this study should understand the risks to any sexual partner of childbearing potential and should practice an effective method of birth control.
* All WOCBP MUST have a negative urine pregnancy test at baseline, or within 7 days prior to receiving investigational product. The minimum sensitivity of the pregnancy test must be 25 IU/L or equivalent units of HCG. If the urine pregnancy test is positive, a serum pregnancy test will then be performed to confirm the result. In the event that both the urine and serum pregnancy tests are positive, the subject must not receive investigational product and must not be enrolled in the study.
* In addition, all WOCBP should be instructed to contact the Investigator immediately if they suspect they might be pregnant (e.g., missed or late menstrual period) at any time during study participation.

The Investigator must immediately notify Amgen in the event of a confirmed pregnancy in a patient participating in the study.

-Prior severe infusion reaction to a human monoclonal antibody.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2007-11 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2016-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ferris, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Ferris RL, Geiger JL, Trivedi S, Schmitt NC, Heron DE, Johnson JT, Kim S, Duvvuri U, Clump DA, Bauman JE, Ohr JP, Gooding WE, Argiris A. Phase II trial of post-operative radiotherapy with concurrent cisplatin plus panitumumab in patients with high-risk, resected head and neck cancer. Ann Oncol. 2016 Dec;27(12):2257-2262. doi: 10.1093/annonc/mdw428. Epub 2016 Oct 11. PMID 27733374

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study included patients with pathologic stage III or IVA squamous cell carcinoma of the oral cavity, larynx, hypopharynx, or human-papillomavirus (HPV) -negative oropharynx, without gross residual tumor, featuring high-risk factors (margins <1mm, extracapsular extension, perineural or angiolymphatic invasion, or ≥2 positive lymph nodes).
Groups:
- Radiation Therapy+Cisplatin+Panitumumab: Postoperative treatment consisted of standard radiation therapy (60-66 Gy over 6-7 weeks) concurrent with weekly cisplatin 30 mg/m^2 and weekly panitumumab 2.5 mg/kg. (no prior chemotherapy, biologic/targeted therapy, or radiation therapy).
Period: Overall Study
Arm/Group | Radiation Therapy+Cisplatin+Panitumumab
Started | 46
Completed | 44
Not Completed | 2
Not completed — Did not receive at least one dose of pan | 2

BASELINE CHARACTERISTICS:
Arm/Group | Radiation Therapy+Cisplatin+Panitumumab
Number analyzed (Participants) | 44
Age, Continuous [Median (Full Range); unit: years] | 58 [23 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 36

OUTCOME MEASURES:

1. Primary Outcome: Probability of Progression-free Survival (PFS) at 2 Years
Time Frame: Up to 90 months for cohort; individual patients up to 24 months after study treatment
Population: Patients who received 60-66 Gy over 6-7 weeks) concurrent with cisplatin 30 mg/m^2 and at least once dose of panitumumab 2.5 mg/kg.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiation Therapy+Cisplatin+Panitumumab
Number analyzed (Participants) | 44
percentage of participants | 70 [58 to 85]

2. Secondary Outcome: Probability of 2-year Overall Survival
Time Frame: Up to 90 months for cohort; individual patients up to 24 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiation Therapy+Cisplatin+Panitumumab
Number analyzed (Participants) | 44
percentage of participants | 72 [60 to 87]

ADVERSE EVENTS:
Arm/Group | Radiation Therapy+Cisplatin+Panitumumab
Serious Adverse Events (participants affected / at risk) | 18/46
Other Adverse Events (participants affected / at risk) | 46/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiation Therapy+Cisplatin+Panitumumab (N=46)
Allergic reaction/hypersensitivity (Immune system disorders) | 1
Anorexia (Gastrointestinal disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 1
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1
Febrile neutropenia (Infections and infestations) | 1
Hemoglobin (Blood and lymphatic system disorders) | 1
Hypotension (Cardiac disorders) | 1
Infection - Other (Specify, __) (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Trachea (Infections and infestations) | 1
Lymphopenia (Blood and lymphatic system disorders) | 3
Mucositis/stomatitis (clinical exam), Oral cavity (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Pain, Chest/thorax NOS (General disorders) | 1
Pain, Pain NOS (General disorders) | 1
Psychosis (hallucinations/delusions) (Nervous system disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Weight loss (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Radiation Therapy+Cisplatin+Panitumumab (N=46)
Auditory/Ear - Other (Specify, __) (Ear and labyrinth disorders) | 3
Tinnitus (Ear and labyrinth disorders) | 3
Platelets (Blood and lymphatic system disorders) | 3
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 3
Lymphopenia (Blood and lymphatic system disorders) | 3
Hemoglobin (Blood and lymphatic system disorders) | 3
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 3
Hypotension (Cardiac disorders) | 3
Hypertension (Cardiac disorders) | 3
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 3
Rigors/chills (General disorders) | 3
Insomnia (General disorders) | 4
Fatigue (asthenia, lethargy, malaise) (General disorders) | 4
Weight loss (General disorders) | 4
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 4
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 4
Ulceration (Skin and subcutaneous tissue disorders) | 4
Wound complication, non-infectious (Skin and subcutaneous tissue disorders) | 4
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4
Pruritus/itching (Skin and subcutaneous tissue disorders) | 4
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 5
Rash: dermatitis associated with radiation, Chemoradiation (Skin and subcutaneous tissue disorders) | 5
Rash: dermatitis associated with radiation, Radiation (Skin and subcutaneous tissue disorders) | 5
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 5
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 6
Gastrointestinal - Other (Specify, __) (Gastrointestinal disorders) | 6
Dehydration (Gastrointestinal disorders) | 6
Diarrhea (Gastrointestinal disorders) | 6
Heartburn/dyspepsia (Gastrointestinal disorders) | 7
Salivary gland changes/saliva (Gastrointestinal disorders) | 7
Anorexia (Gastrointestinal disorders) | 7
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 7
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 7
Mucositis/stomatitis (functional/symptomatic), Oral cavity (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 8
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 8
Mucositis/stomatitis (clinical exam), Oral cavity (Gastrointestinal disorders) | 8
Infection - Other (Specify, __) (Infections and infestations) | 9
Lymphatics - Other (Specify, __) (Blood and lymphatic system disorders) | 9
Edema: head and neck (Blood and lymphatic system disorders) | 10
Creatinine (Metabolism and nutrition disorders) | 10
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 10
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 10
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 11
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 11
Alkaline phosphatase (Metabolism and nutrition disorders) | 11
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 12
Metabolic/Laboratory - Other (Specify, __) (Metabolism and nutrition disorders) | 13
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 14
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 14
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 15
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 15
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 15
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 15
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 16
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 18
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 19
Musculoskeletal/Soft Tissue - Other (Specify, __) (Musculoskeletal and connective tissue disorders) | 22
Mood alteration, Depression (Nervous system disorders) | 22
Dizziness (Nervous system disorders) | 23
Neurology - Other (Specify, __) (Nervous system disorders) | 24
Mood alteration, Anxiety (Nervous system disorders) | 24
Pain, Esophagus (General disorders) | 27
Pain, Pain NOS (General disorders) | 27
Pain, Neck (General disorders) | 29
Pain, Throat/pharynx/larynx (General disorders) | 29
Pain, Oral cavity (General disorders) | 30
Pain - Other (Specify, __) (General disorders) | 30
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 31
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 31
Cough (Respiratory, thoracic and mediastinal disorders) | 35
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes